CLINICAL TRIAL: NCT02767349
Title: Pharmacokinetics and Safety of MNK-155 in Postsurgical Adolescent Subjects With Moderate to Severe Acute Pain
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK15041015
Record Dates: First submitted 2016-04-29; First posted 2016-05-10 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MNK-155 (Experimental): MNK-155, initial dose of two or three tablets followed by 2 tablets every 12 hours up to a maximum of five doses.
  Interventions: Drug: MNK-155

INTERVENTIONS:
Drug: MNK-155 — 2 or 3 tablets initial dose, followed by two tablets every twelve hours

SUMMARY:
An open-label study of the pharmacokinetics (PK) and safety of MNK-155 in postsurgical adolescent subjects aged 12 to 17 years with moderate to severe acute pain. The study will assess the safety of administering multiple doses of MNK-155 in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be male or nonpregnant, nonlactating females between 12 and 17 years of age (inclusive) at time of screening.
2. Subject must have a minimum weight of 100 pounds (45 kg) at the time of screening and have a body mass index (BMI) > 5% and < 95% for their age at the time of screening.
3. Subject must report having moderate or severe acute pain (as determined from the Numerical Pain Rating scale (NPRS) where 0 = no pain, 10 = worst pain; subjects must have a level of 4 or more) after a pediatric surgical procedure (at baseline) that requires hospitalization. Sponsor will pre-approve a list of acceptable surgical procedures prior to study start for each site. Surgical procedures other than those on the pre-approved list may be acceptable on a case by case basis if approved by the medical monitor (MM) and sponsor.
4. Subject, if female of child-bearing potential (defined as postmenarche), must agree to abstain from unprotected sexual activity during study participation and for 2 weeks after study exit/early termination.
5. Subject, if male with reproductive potential, must agree to abstain from unprotected sexual activity during study participation and for 2 weeks after study exit/early termination.
6. Subject, if female of childbearing potential, must have negative pregnancy test (serum or urine) results at screening and check-in.
7. Subject's legally authorized representative (eg, parent, legal guardian) must voluntarily sign and date a parental permission/ Informed Consent that is approved by an Institutional Review Board (IRB), and the subject must sign an IRB approved assent, before undergoing any protocol specific procedures or assessments.
8. Subject and the subject's parent or legal guardian must be able to read, understand, and be willing to follow the study procedures and requirements and communicate meaningfully in English with the investigator and investigator's staff (if the subject cannot read or communicate meaningfully, then the subject's legally authorized representative [eg, parent, legal guardian] must meet this criterion).

Exclusion Criteria:

1. Subject is from a vulnerable population (including mentally disabled children), other than a pediatric population, as defined by the Code of Federal Regulations Title 45, Part 46, Section 46.111(b), including but not limited to employees (temporary, part-time, full time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the clinical research organization, or of the IRB.
2. Subject is expected to require a surgery that could influence the study outcome (eg, ventriculoperitoneal shunt repair in the setting of hydrocephalus).
3. Subject has an abnormal electrocardiogram (ECG) unless the investigator determines the ECG abnormalities are not clinically significant.
4. Subject has a screening pulse oximetry reading of < 95% while awake.
5. Subject has a history of laboratory test results obtained before screening that show the presence of human immunodeficiency virus (HIV), hepatitis B surface antigen, hepatitis C antibody, or active hepatitis A immunoglobulin M.
6. Subject has laboratory values that are greater than 2 times the upper limit of normal (with the exception of white blood cell [WBC] differential values). Enrollment of subjects with laboratory values that are between 1 and 2 times the upper limit of normal (ULN), or below the lower limit of normal, or white blood cells (WBC) differential > 2 x ULN , will be left to the investigator's discretion (no increased risk of participation in study based upon judgment of the investigator).
7. Subject has any history of renal disease that, in the opinion of the investigator, would contraindicate study participation; or subject has significantly impaired renal function, in the opinion of the investigator as evidenced by an estimated glomerular filtration rate calculated using a pediatric appropriate formula such as the Schwartz Equation (Schwartz et al, 2009).
8. Subject has a history or laboratory evidence of bleeding or clotting disorders or conditions.
9. Subject has a known or suspected history of alcoholism, marijuana or illicit drug abuse or misuse within 2 years before screening as evidence from medical history or evidence of tolerance or physical dependence before the first dose of MNK-155.
10. Subject has smoked or used nicotine-containing products within 6 months prior to screening as evidenced by medical history.
11. Subject has a history of psychiatric disorders, such as major depression disorder, anxiety disorders, or psychotic disorders requiring hospitalization and/or medication within 6 months prior to screening. A history of attention deficit hyperactivity disorder requiring medication is acceptable.
12. Subject has a diagnosis of epilepsy or other seizure disorder (a history of febrile seizures is acceptable).
13. Subject has had previous cardiothoracic surgery (subjects who have a history of patent ductus arteriosus ligations/surgery as infants are acceptable).
14. Subject has a history of conditions which might be specifically contraindicated or require caution while using hydrocodone bitartrate (HB), acetaminophen (APAP), and/or ibuprofen (if used as rescue medication) per the Investigator's Brochure (IB) and product information per the appropriate package insert.
15. Subject has a history of any drug allergy, hypersensitivity, or intolerance including HB, APAP, ibuprofen or excipients, or any opioid drug product which, in the opinion of the investigator, would place the subject at particular risk and compromise the safety of the subject in the study.
16. Subject has donated or had significant loss of whole blood (480 mL or more) within 30 days of screening (unless they have received a transfusion and have hematocrit and hemoglobin within the reference range at screening), or plans to donate blood or plasma during the course of the study.
17. Subject has a documented history of any pathologic, iatrogenic or surgical conditions that, in the opinion of the investigator, would compromise the subject's ability to swallow, absorb, metabolize, or excrete MNK-155, including (but not limited to) intractable nausea and/or vomiting, severe GI narrowing, perforation, obstruction, bleed, or gastric band surgery.
18. Subject has a history of a GI event (eg, perforation, obstruction, bleed) within 6 months prior to screening or any GI event greater than 6 months before screening that, in the opinion of the investigator, would make the subject unsuitable for study participation.
19. Subject has received any investigational product or device within 30 days before screening, or is scheduled to receive an investigational device or another investigational drug (other than those in this study) during the course of this study.
20. Subject has used any product containing hydrocodone or APAP within 48 hours prior to the first dose of MNK-155.
21. Subject has a history of conditions which might be specifically contraindicated or require caution to be used during the administration of APAP or HB, including hypersensitivity to HB, or debilitated patients, those with severe impairment of hepatic, pulmonary, or renal function, myxedema or hypothyroidism, adrenocortical insufficiency (Addison's disease), central nervous system (CNS) depression or coma, toxic psychosis, urethral stricture, acute alcoholism, delirium tremens, severe kyphoscoliosis, or biliary tract dysfunction.
22. Subject has any other medical condition, abnormal vital sign (blood pressure, pulse rate, respiratory rate), body temperature, pulse oximetry; or any physical examination or ECG finding at screening which, in the investigator's medical opinion, would preclude safe participation in a clinical study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Time to reach steady state | 12 Hours
Area under the curve | 12 Hours
  Area under the concentration time curves after the first and last dose
Peak exposure | 12 Hours
Half-life | 12 Hours
  Apparent elimination half-life
Time to peak exposure | 12 Hours
  Observed time when peak exposure occurred

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States